CLINICAL TRIAL: NCT04366960
Title: Enoxaparin for Thromboprophylaxis in Hospitalized COVID-19 Patients: Comparison of 40 mg o.d. Versus 40 mg b.i.d. A Randomized Clinical Trial
Brief Title: Comparison of Two Doses of Enoxaparin for Thromboprophylaxis in Hospitalized COVID-19 Patients
Acronym: X-Covid 19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001708-41
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: Open-label Multicentre Prospective Controlled Randomized Trial in patients with SARS-CoV-2 infection. Patients will be randomized 1:1 to 40 mg subcutaneous enoxaparin o.d. versus 40 mg enoxaparin b.i.d within 12 hours after hospitalization.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40 mg subcutaneous enoxaparin o.d. (Active Comparator): Effects of 40 mg subcutaneous enoxaparin o.d.
  Interventions: Drug: Enoxaparin
- 40 mg subcutaneous enoxaparin b.i.d (Active Comparator): Effects of 40 mg subcutaneous enoxaparin b.i.d
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Subcutaneous enoxaparin

SUMMARY:
The purpose of this study is to determine whether a higher dose of low molecular weight heparin (enoxaparin 40 mg b.i.d.) is superior than the standard prophylaxis dose (enoxaparin 40 mg o.d.) in reducing thromboembolic events in COVID-19 patients.

DETAILED DESCRIPTION:
Coronavirus disease-19 (COVID-19 ), which is caused by SARS-CoV-2 infection, are apparently at high risk of venous thromboembolism (VTE), as a consequence of activation of the hemostatic system which, in the most severe cases, can also be associated with the formation of microthrombi and clinically relevant disseminated intravascular coagulation. Concerns about the efficacy of thromboprophylaxis with standard doses of low-molecular-weight heparin (LMWH) has been raised. Therefore, LMWH at higher doses than those recommended for thromboprophylaxis is used in some hospitals, although no evidence exists yet of higher efficacy of high doses compared to standard prophylactic doses. This practice might as well increase the risk of major bleeding. The investigators designed a randomized trial comparing standard prophylactic dose of subcutaneous enoxaparin (40 mg o.d.) with higher dose (40 mg b.i.d) with the aim of testing whether high-dose thromboprophylaxis is more effective than standard dose in preventing VTE in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* All-comers patients aged >=18 years and admitted to hospital with laboratory-confirmed SARS-CoV-2 infection

Exclusion Criteria:

* Patients admitted directly to an intensive care unit;
* Estimated creatinine clearance <15 ml/min/1.73m2;
* Patients needing anticoagulant for prior indication;
* Participants involved in other clinical trials;
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Incidence of venous thromboembolism detected by imaging | 30 days
  Deep vein thrombosis events diagnosed by serial compression ultrasonography and pulmonary embolism events diagnosed by computed tomography scan

SECONDARY OUTCOMES:
In hospital major complications | 30 days
  death, venous thromboembolism, use of mechanical ventilation, stroke, acute myocardial infarction and admission to an intensive care
Number of deep venous thrombosis events | 30 days
  Deep venous thrombosis events diagnosed by serial compression ultrasonography
Sequential organ failure assessment | 30 days
  Maximum sequential organ failure assessment (SOFA) score comparison between the two groups.
  The SOFA score ranges from 0 to 24. Higher SOFA score is associated with a greater risk of death or prolonged intensive care unit stay.
C-reactive protein | 30 days
  To compare C-reactive protein levels as % above the upper reference limit [URL]) among the two groups.
Interleukin-6 | 30 days
  To compare Interleukin-6 levels as % above the upper reference limit [URL]) among the two groups.
D-dimer | 30 days
  To D-dimer compare levels as % above the upper reference limit [URL]) among the two groups.
hs-troponin levels | 30 days
  To compare hs-troponin levels as % above the upper reference limit [URL]) among the two groups.
Acute Respiratory Distress Syndrome | 30 days
  To compare the incidence of SARS-CoV-2-related Acute Respiratory Distress Syndrome (ARDS) between the two groups.
Hospital stay | 30 days
  To compare length of hospital stay between the two groups.
Right ventricular function | 30 days
  To compare measures of right ventricular function at trans-thoracic echocardiography or CT between admission and follow-up, whenever available
Number of pulmonary embolism events | 30 days
  Pulmonary embolism events diagnosed by computed tomography scan

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773
- [Derived] Levi M, Thachil J, Iba T, Levy JH. Coagulation abnormalities and thrombosis in patients with COVID-19. Lancet Haematol. 2020 Jun;7(6):e438-e440. doi: 10.1016/S2352-3026(20)30145-9. Epub 2020 May 11. No abstract available. PMID 32407672